CLINICAL TRIAL: NCT06998264
Title: In-depth Analysis of the Immune Responses in the Upper Respiratory Tract of Influenza-infected Children
Acronym: NoseFlu-Kids
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Arnaud Didierlaurent, Professor, University of Geneva, Switzerland
Other Study IDs: 2024-01409
Record Dates: First submitted 2025-03-28; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Influenza Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasal cells, nasal lining fluid, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Flu kids: Patients aged 2-5 years old hospitalized with flu-like symptoms and a laboratory-confirmed influenza infection

SUMMARY:
The NoseFlu-Kids project aims at characterizing the immune response in the upper respiratory tract in children aged 2 to 5 with a laboratory-confirmed influenza infection. The immune response during the acute phase of the infection and after recovery will be compared to that of control children with no infection or vaccinated with the inactivated flu vaccine by the nasal route (recruited as part of a mirror study in Oxford).

The primary objective of this observational study is to quantify the inflammatory response in the nasal cavity and to correlate it with viral load and with clinical parameters. The study also aims to compare the inflammatory response measured in the nose to that measured in the blood.

Participants will have two study visits including a blood draw, several nasal samplings (nasal lining fluid and nasal cells) and a saliva sampling, one within 72 hours of their hospital admission and another one month later. Nasal lining fluid and saliva will be obtained every two or three days until symptoms disappear. During those visits, questions regarding symptoms will be asked.

ELIGIBILITY:
Inclusion criteria:

* Aged 2-5 years
* Presenting clinical signs of an influenza-like illness
* Having a concomitant positive laboratory test for influenza.

Exclusion criteria:

* Immunosuppression
* Intubation or under invasive mechanical ventilation
* Co-infection with RSV or SARS-CoV-2

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited among patients hospitalized or visiting the emergencies at the Geneva University Hospitals (HUG).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pro-inflammatory cytokine levels in nasal fluid by a multiplex assay | 1 month

SECONDARY OUTCOMES:
Phenotypes and frequencies of immune in nasal cavity and in blood cells by flow cytometry | 1 month
Influenza-specific antibody titers in nasal fluid and blood by ELISA or multiplex assay | 1 month
Influenza virus load by specific quantitative RT-PCR assay in nasal cavity and/or saliva | 1 month
Levels of blood cytokines by multiplex assay | 1 month
Clinical outcome measure 1: nature and severity of symptoms | 1 month
Clinical outcome measure 2: number of days with fever | 1 month
Clinical outcome measure 3: number of days with oxygen | 1 month
Clinical outcome measure 4: highest FiO2 | 1 month
Clinical outcome measure 5: secondary bacterial infection | 1 month
Clinical outcome measure 6: transfer to ICU or IMCU | 1 month
Clinical outcome measure 7: length of stay in intensive care | 1 month
Clinical outcome measure 8: intubation or mechanical ventilation | 1 month
Clinical outcome measure 9: mortality | 1 month
Clinical outcome measure 10: rehospitalization | 1 month
Clinical outcome measure 11: medical consultation for a respiratory disease | 1 month
Clinical outcome measure 12: new prescription of antibiotics or corticosteroids | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Didierlaurent, PhD, Principal Investigator — University of Geneva; Arnaud L'Huillier, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland